CLINICAL TRIAL: NCT04048161
Title: Study of Tacrolimus vs Mycophenolate Mofetil in Pediatric Patients With Frequently Relapsing or Steroid Dependent Nephrotic Syndrome: a Randomized, Multicenter, Open-label, Parallel-arm Study
Brief Title: Study of Tacrolimus vs Mycophenolate Mofetil in Pediatric Patients With Nephrotic Syndrome
Acronym: STAMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Children's Hospital of Fudan University (Other); Peking University First Hospital (Other); First Affiliated Hospital of Zhongshan Medical University (Other); Nanjing Children's Hospital (Other); Chengdu Women and Children's Center Hospital (Other); Tongji Hospital (Other); Second Xiangya Hospital of Central South University (Other); Children's Hospital of Chongqing Medical University (Other); Children's Hospital of Soochow University (Other); Henan Provincial People's Hospital (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Mao Jianhua, Chief Physician, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAMP
Record Dates: First submitted 2019-07-30; First posted 2019-08-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Nephrotic Syndrome in Children
Keywords: Nephrotic Syndrome; Frequently Relapsing Nephrotic Syndrome; Steroid Dependent Nephrotic Syndrome; Tacrolimus; Mycophenolate mofetil
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus(Group A) (Experimental): Tacrolimus: 0.5mg and 1mg; Capsule; 0.05-0.10mg/kg/day，BID; Steroid: 5mg; Oral tablets; 1.0-1.5 mg/kg, qod or 0.5-0.75 mg/kg/day, qd;
  Interventions: Drug: Tacrolimus
- Mycophenolate Mofetil(Group B) (Active Comparator): Mycophenolate Mofetil: 250mg; Dispersible tablets; 20~30mg/kg/day，BID; Steroid: 5mg; Oral tablets; 1.0-1.5 mg/kg, qod or 0.5-0.75 mg/kg/day, qd;
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Tacrolimus — The patients will be divided into two groups randomly. Tacrolimus dose: 0.05-0.10 mg/kg/day, BID. The concentration for tacrolimus is 5-10 ng/ml，then reduce the dosage of drugs to maintian the concentration for tacrolimus is < 5ng/ml. Total duration : 1 year.
  Steroid dose: 1.0-1.5 mg/kg, qod or 0.5-0.75 mg/kg/day, qd， then gradually taper the steroid to 5mg/day.
  Other Names: Tacrolimus capsules（CYONSE®）
  Arms: Tacrolimus(Group A)
Drug: Mycophenolate Mofetil — The patients will be divided into two groups randomly. Mycophenolate Mofetil dose: 20~30mg/kg/day，BID. The concentration for MPA-AUC is 30~50 μg.h/ml，then reduce the dosage of drugs to maintian the concentration for MPA-AUC is ≤40 μg.h/ml. Total duration : 1 year.
  Steroid dose: 1.0-1.5 mg/kg, qod or 0.5-0.75 mg/kg/day, qd， then gradually taper the steroid to 5mg/day.
  Other Names: Mycophenolate Mofetil Dispersible tablets（CYCOPIN®）
  Arms: Mycophenolate Mofetil(Group B)

SUMMARY:
Primary nephrotic syndrome accounts for approximately 90% of the total number of nephrotic syndrome in childhood and it is the most common glomerular disease in children. Although treatment with steroids is uesful for primary nephrotic syndrome, proning to cause frequent relapse/steroid-dependent nephrotic syndrome after treatment, and the usage of immunosuppressive agents has become a new choice for the treatment of such patients. This study is a prospective, randomized, multicenter, open, parallel controlled trial, evaluating the efficacy and safety of steroid combined with the immunosuppressive agents which are tacrolimus and mycophenolate mofetil to children who with frequently relapsing or steroid-dependent nephrotic syndrome, all we wish to obtain the proper drug choice and individualized treatment options for children with nephrotic syndrome.

DETAILED DESCRIPTION:
Although steroids are recognized as first-line treatments for nephrotic syndrome, the vast majority of children relapse, and about half of them have frequent relapse or steroids dependence after treatment with steroids alone. Some children experienced steroids-resistance after multiple relapses, and eventually developed into chronic kidney dysfunction. Long-term or repeated application of large doses of steroids will lead to side effects such as obesity, growth retardation, and hypertension. Although the treatment of steroids with immunosuppressive agents is a new choice for the treatment of such patients, traditional immunosuppressive agents such as cyclophosphamide and cyclosporine A will bring some serious irreversible side effects, while immunosuppressive agents tacrolimus has the dual effects of immunosuppression and podocyte protection, and is more widely used in the department of nephrology, what's more, the other immunosuppressive agents mycophenolate mofetil has advantage of no kidney toxic, less adverse reactions and higher safety, which gradually being valued by nephrologists in recent years. This study mainly compares the efficacy and safety of tacrolimus and mycophenolate mofetil in the treatment of children with frequently relapsing or steroids-dependent nephrotic syndrome, in order to provide a more effective and safer treatment for children with nephrotic syndrome as well as the therapeutic medication options.

ELIGIBILITY:
Inclusion Criteria:

* Sensitive but frequent relapses or steroids dependence nephrotic syndrome
* Age: 2 to 18 years old
* Normal renal function: estimated glomerular filtration rate ≥90ml/min/1.73m2
* Morning urine protein <1+ or urine protein-creatinine ratio <0.2g/g (<20 mg/mmol) for 3 consecutive days and above when in enroll
* No tacrolimus, mycophenolate mofetil, cyclosporine A, rituximab or cyclophosphamide was used within 2 years prior to the enrollment

Exclusion Criteria:

* steroids-resistant nephrotic syndrome
* Family history of nephrotic syndrome, chronic glomerulonephritis or uremia
* Leukopenia (White Blood Cells ≤ 3.0 * 10^9 / L)
* Moderate to severe anemia (hemoglobin <9.0 g/dL)
* Thrombocytopenia (platelet count <100*10^12/L)
* Positive Hepatitis B virus serological indicators (Hepatitis B surface antigen or / and Hepatitis B virus e antigen or / and Hepatitis B core antibody), Hepatitis C virus-positive or patients with abnormal liver function (2 or more times of alamine aminotransferase or total bilirubin was exceeded the normal value, and continued to rise for 2 weeks)
* There are chronic active infections such as Epstein-Barrvirus, cytomegalovirus or Mycobacterium tuberculosis, and the usage of steroids and immunosuppressive agents may aggravate the state of an illness
* Secondary nephrotic syndrome (such as purpuric nephritis, lupus nephritis, etc.)
* Those who with hematological or endocrine system diseases as well as serious organs illness such as heart, liver or kidney
* Those who with other autoimmune diseases or primary immunodeficiencies or tumors
* Those who was known to be sensitized to tacrolimus, mycophenolate mofetil, glucocorticoids, or any of the above drugs
* Those who have participated in other clinical trials within three months prior to the enrollment
* Those who was not suitable for participating this study judged by investigator

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
1-year relapse-free survival rate | 1-year period after randomization
  The rate of no relapse within 1 year

SECONDARY OUTCOMES:
Relapse of nephrotic syndrome during 12 months after randomization | 1-year period after randomization
  Proportion of patients with one or more relapse(s) of nephrotic syndrome
Number of relapses during 12 months follow up | 1-year period after randomization
  Number of nephrotic syndrome relapses per patient year during the 12 months period after randomization
The first time to relapse | 1-year period after randomization
  The first time to relapse after patients taking part in this study
Cumulative prednisone dosage (milligrams per kilogram per year) | 1-year period after randomization
  The total dosage of prednisones from the beginning to the end of the trial
Change in serum cholesterol, hemoglobin and blood albumin of the patients | 1-year period after randomization
  The changes of serum cholesterol, hemoglobin and blood albumin in each follow-up during the study
Change in renal function of the patients | 1-year period after randomization
  The change for renal function was judged by the changes of serum creatinine and estimated glomerular filtration rate in each follow-up during the study
Change in anthropometry and growth velocity during 12-month period after randomization | 1-year period after randomization
  Changes in standard deviation scores for weight, height and body mass index during 12-month period after randomization
Adverse event | 1-year period after randomization
  The number of harmful reactions and the types of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, MD, Study Chair — Children's Hospital, Zhejiang University School of Medicine
Locations (12):
- China (12):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Zhongshan Medical University, Guangzhou, Guangdong
  - Henan Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Shandong Provincial Hospital, Jinan, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Women and Children's Center Hospital, Chengdu, Shichuan
  - The Children Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
We could not share data without patients' agreement.

REFERENCES:
- [Result] Ren H, Shen P, Li X, Pan X, Zhang W, Chen N. Tacrolimus versus cyclophosphamide in steroid-dependent or steroid-resistant focal segmental glomerulosclerosis: a randomized controlled trial. Am J Nephrol. 2013;37(1):84-90. doi: 10.1159/000346256. Epub 2013 Jan 22. PMID 23343906
- [Result] Filler G, Young E, Geier P, Carpenter B, Drukker A, Feber J. Is there really an increase in non-minimal change nephrotic syndrome in children? Am J Kidney Dis. 2003 Dec;42(6):1107-13. doi: 10.1053/j.ajkd.2003.08.010. PMID 14655180
- [Result] Eddy AA, Symons JM. Nephrotic syndrome in childhood. Lancet. 2003 Aug 23;362(9384):629-39. doi: 10.1016/S0140-6736(03)14184-0. PMID 12944064
- [Result] Wong W. Idiopathic nephrotic syndrome in New Zealand children, demographic, clinical features, initial management and outcome after twelve-month follow-up: results of a three-year national surveillance study. J Paediatr Child Health. 2007 May;43(5):337-41. doi: 10.1111/j.1440-1754.2007.01077.x. PMID 17489822
- [Result] Tarshish P, Tobin JN, Bernstein J, Edelmann CM Jr. Prognostic significance of the early course of minimal change nephrotic syndrome: report of the International Study of Kidney Disease in Children. J Am Soc Nephrol. 1997 May;8(5):769-76. doi: 10.1681/ASN.V85769. PMID 9176846
- [Result] Shaw KT, Ho AM, Raghavan A, Kim J, Jain J, Park J, Sharma S, Rao A, Hogan PG. Immunosuppressive drugs prevent a rapid dephosphorylation of transcription factor NFAT1 in stimulated immune cells. Proc Natl Acad Sci U S A. 1995 Nov 21;92(24):11205-9. doi: 10.1073/pnas.92.24.11205. PMID 7479966
- [Result] Koefoed-Nielsen PB, Karamperis N, Hojskov C, Poulsen JH, Jorgensen KA. The calcineurin activity profiles of cyclosporin and tacrolimus are different in stable renal transplant patients. Transpl Int. 2006 Oct;19(10):821-7. doi: 10.1111/j.1432-2277.2006.00359.x. PMID 16961774
- [Result] Neidle S, Goodwin GH. A homology-based molecular model of the proline-rich homeodomain protein Prh, from haematopoietic cells. FEBS Lett. 1994 May 30;345(2-3):93-8. doi: 10.1016/0014-5793(94)00446-3. PMID 7911091
- [Result] Sepe V, Libetta C, Giuliano MG, Adamo G, Dal Canton A. Mycophenolate mofetil in primary glomerulopathies. Kidney Int. 2008 Jan;73(2):154-62. doi: 10.1038/sj.ki.5002653. Epub 2007 Nov 7. PMID 17989649
- [Result] Briggs WA, Choi MJ, Scheel PJ Jr. Successful mycophenolate mofetil treatment of glomerular disease. Am J Kidney Dis. 1998 Feb;31(2):213-7. doi: 10.1053/ajkd.1998.v31.pm9469489.
- [Result] Gellermann J, Weber L, Pape L, Tonshoff B, Hoyer P, Querfeld U; Gesellschaft fur Padiatrische Nephrologie (GPN). Mycophenolate mofetil versus cyclosporin A in children with frequently relapsing nephrotic syndrome. J Am Soc Nephrol. 2013 Oct;24(10):1689-97. doi: 10.1681/ASN.2012121200. Epub 2013 Jun 27. PMID 23813218
- [Result] Schwartz GJ, Brion LP, Spitzer A. The use of plasma creatinine concentration for estimating glomerular filtration rate in infants, children, and adolescents. Pediatr Clin North Am. 1987 Jun;34(3):571-90. doi: 10.1016/s0031-3955(16)36251-4. PMID 3588043
- [Derived] Wang J, Liu F, Yan W, Zhou J, Zhang Y, Rong L, Jiang X, Zhao F, Zhu C, Wu X, Li X, Sun S, Wang J, Wang M, Yang Q, Xu H, Chen J, Liu C, Tian M, Feng S, Duan Q, Zhong X, Zhu Y, Li X, Fu H, Huang L, Ma D, Ding J, Ye Q, Mao J. Tacrolimus or Mycophenolate Mofetil for Frequently Relapsing or Steroid-Dependent Nephrotic Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2025 May 12;179(7):722-9. doi: 10.1001/jamapediatrics.2025.0765. Online ahead of print. PMID 40354041
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526

DOCUMENTS (2):
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT04048161/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT04048161/SAP_001.pdf